CLINICAL TRIAL: NCT07284654
Title: A Phase 3, Randomized, Double-Blind, Active-Controlled Clinical Study to Evaluate the Safety, Tolerability, and Immunogenicity of VAX-31 in Healthy Subjects 50 Years of Age and Older With Immunobridging to Subjects 18-49 Years of Age
Brief Title: Safety, Tolerability, and Immunogenicity of VAX-31 in Adults ≥50 Years With Immunobridging to Adults 18-49
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Vaxcyte, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VAX31-103
Record Dates: First submitted 2025-12-08; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Pneumococcal Vaccines
Keywords: 31 Valent PCV; Pneumonia; Pneumococcal Infection
MeSH Terms: conditions — Pneumonia; Pneumococcal Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1 (VAX-31), participant ≥ 50 years of age (Experimental): Participants will receive a single dose of VAX-31 administered via intramuscular injection at Day 1
  Interventions: Biological: 31 valent pneumococcal conjugate vaccine
- Cohort 1 (PCV21), participant ≥ 50 years of age (Active Comparator): Participants will receive a single dose of PCV21 (Capvaxive) administered via intramuscular injection at Day 1
  Interventions: Biological: PCV21
- Cohort 1 (PCV20), participant ≥ 50 years of age (Active Comparator): Participants will receive a single dose of PCV20 (Prevnar 20) administered via intramuscular injection at Day 1
  Interventions: Biological: PCV20
- Cohort 2 (VAX-31), participant 18-49 years of age (Experimental): Participants will receive a single dose of VAX-31 administered via intramuscular injection at Day 1
  Interventions: Biological: 31 valent pneumococcal conjugate vaccine
- Cohort 2 (PCV20), participant 18-49 years of age (Active Comparator): Participants will receive a single dose of PCV20 (Prevnar 20) administered via intramuscular injection at Day 1
  Interventions: Biological: PCV20

INTERVENTIONS:
Biological: 31 valent pneumococcal conjugate vaccine — 0.5 mL of VAX-31 will be administered into the deltoid muscle
  Arms: Cohort 1 (VAX-31), participant ≥ 50 years of age; Cohort 2 (VAX-31), participant 18-49 years of age
Biological: PCV20 — 0.5 mL of the 20 valent pneumococcal conjugate vaccine will be administered into the deltoid muscle
  Other Names: Prevnar 20
  Arms: Cohort 1 (PCV20), participant ≥ 50 years of age; Cohort 2 (PCV20), participant 18-49 years of age
Biological: PCV21 — 0.5 mL of the 21 valent pneumococcal conjugate vaccine will be administered into the deltoid muscle
  Other Names: Capvaxive
  Arms: Cohort 1 (PCV21), participant ≥ 50 years of age

SUMMARY:
The primary objectives of this study are to evaluate the safety, tolerability, immunologic noninferiority (for shared serotypes) and immunologic superiority (for novel serotypes) of VAX-31 compared to PCV21 and PCV20 in adults ≥50 years of age, and to bridge the immune responses induced by VAX-31 in adults 50-64 years of age to adults 18-49 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥18 years of age (inclusive) at the time of randomization into the study.
* Able and willing to complete the informed consent process.
* Available for clinical follow-up through the last study visit.
* In good general health or with stable underlying chronic condition(s), as determined by medical history, oral temperature, physical examination, and clinical judgment of the Investigator (ongoing chronic conditions must be documented as stable per Investigator).
* Willing to have blood samples collected and used for research purposes.
* Able to provide proof of identity to the satisfaction of the site personnel completing the enrollment process.
* Female participants of childbearing potential, defined as premenopausal females capable of becoming pregnant, must have a negative urine pregnancy test immediately prior to randomization and agree to use acceptable contraception. Male subjects with partners of childbearing potential must agree to practice an acceptable contraception method.
* Able to access and use a device connected to Wi-Fi or cellular network for completion of an electronic diary (eDiary).

Exclusion Criteria:

* History of invasive pneumococcal disease (IPD) or pneumococcal pneumonia (either confirmed or self-reported) at any age.
* Previous receipt of any licensed or investigational pneumococcal vaccine at any age.
* Receipt of any investigational product within 30 days prior to Day 1, currently participating in another interventional investigational study, or having plans to receive another investigational product(s) while on study.
* Receipt of any live vaccine within 30 days prior to Day 1, or receipt of any non-live (including inactivated) vaccine within 14 days prior to Day 1.
* Body temperature >38.0°C (>100.4°F) or acute illness within 3 days prior to study vaccination (subject may be rescreened).
* Current diagnosis of human immunodeficiency virus, Hepatitis B, or Hepatitis C.
* History of severe allergic reaction with generalized urticaria, angioedema, or anaphylaxis to any previous vaccination.
* Individual who is pregnant, breastfeeding, or planning to become pregnant during study participation.
* Has a known or suspected immunocompromising condition, including, but not limited to, leukemia, lymphoma, chronic renal failure, or congenital or acquired immunodeficiency.
* Bleeding disorder diagnosed by a doctor (e.g., factor deficiency, coagulopathy, or platelet disorder requiring special precautions) resulting in clinically significant bruising or bleeding difficulties with IM injections or blood draws.
* Receipt of blood or blood product (including polyclonal intravenous immunoglobulin) within 60 days prior to enrollment into the study.
* Is currently receiving immunosuppressive or immune-modifying therapy, including systemic corticosteroids (this includes ≥3 months of prednisone equivalent from 5 to <10 mg/day and ≥2 weeks of prednisone equivalent ≥10 mg/day).
* Received any part of a ≥14-day course of systemic corticosteroids (prednisone equivalent >10 mg/day) within 14 days of study vaccination.
* History of malignancy ≤5 years before enrollment, except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer.
* Any medical, psychiatric, or social condition that in the judgment of the Investigator is a contraindication to protocol participation or impairs a subject's ability to give informed consent.
* Employee of, or first-degree relative of, any person employed by the Sponsor, the contract research organization (CRO), the Investigator, site personnel, or site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4000 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Serotype-specific OPA geometric mean titers (GMT) in 50 year olds and above | 1 month after vaccination
Percentage of subjects reporting solicited local adverse events (AE) (redness, swelling, and pain at injection site) | up to 7 days after vaccination
Percentage of subjects reporting solicited systemic AE (fever, headache, fatigue, muscle pain, and joint pain) | up to 7 days after vaccination
Percentage of subjects reporting unsolicited AE | up to 31 days after vaccination
Percentage of subjects reporting serious adverse events (SAE), new onset of chronic illness (NOCI), and medically attended adverse events (MAAE) | up to 6 Months after vaccination
Serotype-specific OPA geometric mean titers (GMT) in 18 to 49 year olds and 50 to 64 year olds | 1 month after vaccination

SECONDARY OUTCOMES:
Serotype-specific IgG geometric mean concentrations (GMC) in 50 year olds and above | 1 month after vaccination
Serotype-specific IgG GMC in 18 to 49 year olds and 50 to 64 year olds | 1 month after vaccination

CONTACTS AND LOCATIONS:
Locations (30):
- United States (30):
  - Accel Research Site - Achieve - Birmingham - ERN, Birmingham, Alabama
  - Center for Indigenous Health - Chinle - Johns Hopkins Project, Chinle, Arizona
  - Center for Indigineous Health - Whiteriver - John Hopkins Project, Whiteriver, Arizona
  - Clinical Innovations Trials - Riverside - CenExel, Riverside, California
  - Research Centers of America - Hollywood - CenExel, Hollywood, Florida
  - Health Awareness - Jupiter - ERN, Jupiter, Florida
  - Suncoast Research Group LLC, Miami, Florida
  - Precision Clinical Research - Sunrise, Sunrise, Florida
  - Clinical Research Atlanta - Headlands, Stockbridge, Georgia
  - Velocity Clinical Research - Valparaiso (Buynak Clinical Research), Valparaiso, Indiana
  - Johnson County Clin-Trials - JCCT, Lenexa, Kansas
  - Alliance for Multispecialty Research, LLC - West Wichita, Wichita, Kansas
  - DelRicht Clinical Research, LLC - New Orleans, New Orleans, Louisiana
  - Headlands Research - Detroit - Headlands, Southfield, Michigan
  - DelRicht Research, LLC - Gulfport, Gulfport, Mississippi
  - Sky Integrative Medical Center - SKYCRNG, Ridgeland, Mississippi
  - Alliance for Multispecialty Research, LLC - Kansas City, Kansas City, Missouri
  - Velocity Clinical Research, Omaha, Nebraska
  - Advanced Memory Research Institute - CenExe, Toms River, New Jersey
  - Center for Indigineous Health - Gallup - John Hopkins Project, Gallup, New Mexico
  - Center for Indigineous Health - Shiprock - John Hopkins Project, Shiprock, New Mexico
  - Rochester Clinical Research - ATLAS - Rochester, Rochester, New York
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Lynn Institute of Norman, Norman, Oklahoma
  - DM Clinical Research - Philadelphia, Philadelphia, Pennsylvania
  - Coastal Carolina Research Center - Alcanza - HyperCore, North Charleston, South Carolina
  - Flourish Research - San Antonio, San Antonio, Texas
  - DM Clinical Research - Sugarland, Sugar Land, Texas
  - JBR Clinical Research - CenExel JBR, Salt Lake City, Utah
  - Charlottesville Medical Research Center - Alcanza - HyperCore, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Vaxcyte is committed to providing access to anonymized data from the company's clinical trials for the purpose of legitimate scientific research. Requests for data may be addressed to datasharing@vaxcyte.com. Requests must be accompanied by a detailed analysis plan and will be reviewed for scientific validity. Data will be made available after initial product approval. Sharing of data may require execution of a data-sharing agreement.
Supporting Information: Study Protocol
Time Frame: Individual participant data will be shared after deidentification and made available starting 6 months after initial product approval.
Access Criteria: Criteria will depend on the specific proposal received and may include qualification of the scientific researchers, potential contribution to the research field, scientific rigor of statistical and analytical methods, and other criteria appropriate for the proposal.